CLINICAL TRIAL: NCT06445075
Title: A Phase 2 Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Efficacy, Safety and Pharmacokinetics of Apitegromab in Overweight and Obese Adult Subjects
Brief Title: Efficacy and Safety of Apitegromab for the Treatment of Adults Who Are Overweight or Obese
Acronym: EMBRAZE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Scholar Rock, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SRK-015-006
Record Dates: First submitted 2024-05-22; First posted 2024-06-06 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Overweight and Obesity
Keywords: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — apitegromab; Tirzepatide

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Active treatment, randomized, double-blind, placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Apitegromab + incretin mimetic
  Interventions: Drug: Apitegromab; Drug: Tirzepatide
- Cohort 2 (Placebo Comparator): Placebo + incretin mimetic
  Interventions: Drug: Placebo; Drug: Tirzepatide

INTERVENTIONS:
Drug: Apitegromab — Apitegromab (SRK-015) is a fully human anti-proMyostatin monoclonal antibody (mAb) that specifically binds to human pro/latent myostatin, inhibiting myostatin activation. Apitegromab was administered every 4 weeks by intravenous (IV) infusion.
  Other Names: SRK-015
  Arms: Cohort 1
Drug: Placebo — Same appearance and composition as apitegromab drug product but does not contain the active ingredient. Placebo was administered every 4 weeks by intravenous (IV) infusion.
  Arms: Cohort 2
Drug: Tirzepatide — Glucose-dependent insulinotropic polypeptide (GIP) receptor and glucagon-like peptide-1 (GLP-1) receptor agonist. Tirzepatide was administered every week by subcutaneous injection.
  Other Names: ZEPBOUND

SUMMARY:
A phase 2 study to evaluate the effects of apitegromab as an adjunctive therapy to GLP-1 receptor agonist therapy in subjects with overweight or obesity

DETAILED DESCRIPTION:
This phase 2 randomized, double-blind, placebo-controlled, multicenter study assessed the safety, efficacy, and pharmacokinetics (PK) of apitegromab when used as an adjunctive therapy to GLP-1 receptor agonist therapy in subjects with overweight and obesity and without diabetes. Each subject received tirzepatide throughout the treatment period. In addition, all subjects were randomized 1:1 to receive either apitegromab or placebo during the treatment period.

ELIGIBILITY:
Inclusion Criteria

* Able to comprehend the informed consent process and provide written informed consent prior to study enrollment and the conduct of any study-related assessments to study enrollment and the conduct of any study-related assessments
* Male or female, age ≥ 18 and ≤ 65 years at the time of informed consent
* Stable body weight (±5 kg) within 90 days of Screening
* At Screening, a BMI of:

  1. ≥30.0 kg/m2 to ≤45.0 kg/m2 or
  2. ≥27.0 kg/m2 to <30.0 kg/m2 with the presence of 1 or more weight-related comorbid condition(s). Note: See exclusion criteria for specific organ class disease parameters

Exclusion Criteria:

* History of or active cardiovascular, neurovascular, peripheral vascular, pulmonary, hepatic, pancreatic, neuromuscular, and/or psychiatric disease
* Active malignancy, other than local subcutaneous squamous cell and basal cell carcinomas
* History of immunosuppressive, chemotherapeutic, or radiation treatment within 12 months prior to Screening
* History of Type 1 diabetes or active Type 2 diabetes (T2D). If there was a history of T2D and it resolved, then the resolution must have occurred >12 months prior to Screening. Prediabetes managed with nonpharmacologic approaches (exercise and diet) is not an exclusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2024-05-21 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-06-17 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in total Lean Body Mass (kg) at 24 weeks | Baseline and 24 weeks
  Dual-energy X-ray absorptiometry was used to evaluate body composition

SECONDARY OUTCOMES:
Change from Baseline in body weight | Baseline and 24 weeks
  Total body weight was assessed via a calibrated scale
Change from Baseline in percent lean body mass (%) | Baseline and 24 weeks
  Dual-energy X-ray absorptiometry was used to evaluate body composition
Change from Baseline in fat body mass (kg and %) | Baseline and 24 weeks
  Dual-energy X-ray absorptiometry was used to evaluate body composition
Change from Baseline in visceral adipose tissue (VAT), subcutaneous adipose tissue (SAT), and trunk fat body mass (kg and %) | Baseline and 24 weeks
  Dual-energy X-ray absorptiometry was used to evaluate body composition
Percent (%) of weight loss from baseline due to fat body mass loss | Baseline and 24 weeks
  Dual-energy X-ray absorptiometry was used to evaluate body composition
Percent (%) of weight loss from baseline due to lean body mass loss | Baseline and 24 weeks
  Dual-energy X-ray absorptiometry was used to evaluate body composition
Concentration of apitegromab in circulation over time | Baseline up to 40 weeks
  Blood samples were assessed for circulating concentration of apitegromab
Concentration of latent myostatin in circulation over time | Baseline up to 24 weeks
  Blood samples were assessed for circulating concentration of latent myostatin
Treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) | Baseline up to 40 weeks
  Incidence and severity of TEAEs and SAEs
Presence of anti-drug antibodies (ADA) against apitegromab over time | Baseline up to 40 weeks
  Measured in serum blood samples

OTHER OUTCOMES:
Change from Baseline in HbA1c | Baseline up to 32 weeks
  Blood samples were assessed for HbA1c (glycated hemoglobin)
Change from baseline in fasting serum triglycerides | Baseline up to 32 weeks
  Blood samples were assessed for fasting serum triglycerides
Change from baseline in total cholesterol | Baseline up to 32 weeks
  Blood samples were assessed for total cholesterol
Change from baseline in low-density lipoprotein cholesterol (LDL-C) | Baseline up to 32 weeks
  Blood samples were assessed for low-density lipoprotein cholesterol (LDL-C)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - ProSciento CRU, Chula Vista, California
  - AdventHealth Translational Research Institute, Orlando, Florida
  - Great Lakes Clinical Trials, LLC d/b/a Flourish Research, Chicago, Illinois
  - Tandem Clinical Research GI, LLC, Marrero, Louisiana
  - Alliance for Multispecialty Research, LLC, Norman, Oklahoma
  - Apex Mobile Clinical Research, Bellaire, Texas
  - Clinical Trials of Texas, LLC dba Flourish Research, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes